CLINICAL TRIAL: NCT03710824
Title: Investigating Trends in Quality of Life in Patients With Idiopathic Pulmonary Fibrosis (IPF) Under Treatment With Nintedanib
Acronym: QUALIFY IPF
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0355
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Nintedanib for patients with Idiopathic Pulmonary Fibrosis
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — diagnosed IPF patients initiating treatment with nintedanib

SUMMARY:
Multi-center, non-interventional, prospective cohort study aiming to enroll 240 Idiopathic Pulmonary Fibrosis patients receiving treatment with nintedanib in a consecutive manner from 10-12 reference centers across Greece.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥40 years of age.
* Patients that have signed Informed Consent Form.
* Treatment naive patients with an initial IPF diagnosis no more than 3 months prior to enrolment according to 2011 American Thoracic Society (ATS)/ European Respiratory Society (ERS)/ Japanese Respiratory Society (JRS)/Latin American Thoracic Association (ALAT) guidelines who are initiating treatment with nintedanib (as monotherapy for IPF) the latest on the enrollement day or have initiated treatment with nintedanib (as monotherapy for IPF) within the past 7 days prior to enrolment.
* Patients for whom the decision to prescribe therapy with nintedanib according to the locally approved product's Summary of Product Characteristics (SmPC) has already been taken prior to their enrolment in the study and is clearly separated from the physician's decision to include the patient in the current study.
* Patients that are able to read, understand and complete the study specific questionnaires.

Exclusion Criteria:

* Treatment with nintedanib for more than 7 days prior to study enrolment.
* Patients receiving a combination therapy of nintedanib & pirfenidone for IPF.
* Patients that meet any of the contraindications to the administration of the study drug nintedanib according to the approved SmPC.
* Prior treatment with pirfenidone or other treatment for IPF.
* Participation in an interventional study.
* Patients currently receive treatment with any investigational drug/device/intervention or have received any investigational product within 1 month or 5 half-lives of the investigational agent (whichever is longer) before the initiation of therapy with nintedanib.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed IPF patients initiating treatment with nintedanib according to their physician's clinical decision will be enrolled in this study. In details, patients will be eligible to enroll in the study if the fulfil all the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Greece (10):
  - University General Hospital of Evros, Alexandroupoli
  - Gen. Hosp. of Chest Diseases "Sotiria", Univ. Resp. Med., Athens
  - University General Hospital Attikon, Athens
  - General Hospital of Kerkyra, Corfu
  - University Hospital of Heraklion, University Pulmonology Cl, Heraklion
  - Univ. Gen. Hosp. of Ioannina, Ioannina
  - General University Hospital of Larissa, Larissa
  - Univ. Gen. Hosp. of Patras, Pátrai
  - A Pulmonology Clinic "G.Papanikolaou" Hospital Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This observational study aimed to collect data on various patient reported outcomes (PROs) in patients with idiopathic pulmonary fibrosis (IPF) under treatment with nintedanib (QUALIFY Idiopathic Pulmonary Fibrosis) over a 52-week period in Greece. Data of 180 newly diagnosed IPF patients enrolled from 10 University Pulmonology Clinics and Reference Centers of the Public Hospital Setting were collected.
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the clinical trial at any time for any reason given. Close monitoring of all subjects was adhered to throughout the trial conduct. Treatment interruption and dose reduction were allowed as medically indicated. Rescue medication was allowed for all subjects as required.
Groups:
- Nintedanib for Patients With Idiopathic Pulmonary Fibrosis: Patients were considered eligible if they were ≥40 years old y/o, had signed informed consent form, were treatment-naïve with an initial IPF diagnosis no more than 3 months prior to enrolment and were initiating treatment with nintedanib (as monotherapy) the latest on the enrolment day or had initiated it within the past 7 days prior to enrolment, and for whom the decision to prescribe treatment with nintedanib was according to the locally approved treatment label.
Period: Overall Study
Arm/Group | Nintedanib for Patients With Idiopathic Pulmonary Fibrosis
Started | 180
Completed | 149
Not Completed | 31
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 25
Not completed — Treatment discontinuation | 2

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): all patients who were enrolled in the trial and have received at least once nintedanib during the trial. Any analysis on primary, secondary and safety endpoints was performed in the TS.
Arm/Group | Nintedanib for Patients With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 180
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.96 (7.829)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 136
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 180
  More than one race | 0
  Unknown or Not Reported | 0
St. George's Respiratory Questionnaire (SGRQ) scores at baseline [Mean (Standard Deviation); unit: Score on a scale] — SGRQ is a 50-item questionnaire assessing 3 domains: symptoms (frequency and severity of respiratory symptoms), activity (activities that cause, or are limited by, breathlessness) and psychosocial impact (range of aspects concerning social functioning and the psychological impact of the disease) that was self-completed by patients at all study visits. The total SGRQ score and the score for each domain range from 0 to 100, with higher scores indicating worse HRQoL.
  Score on a scale
    SGRQ total score | 32.93 (19.319)
    symptom domain score | 32.09 (21.089)
    activity domain score | 48.19 (22.956)
    psychosocial impact score | 24.01 (20.487)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Health Related Quality of Life (HRQoL) Using SGRQ Score at 3 Months
Description: St. George's Respiratory Questionnaire (SGRQ) is a 50-item questionnaire assessing 3 domains: symptoms (frequency and severity of respiratory symptoms), activity (activities that cause, or are limited by, breathlessness) and psychosocial impact (range of aspects concerning social functioning and the psychological impact of the disease) that was self-completed by patients at all study visits. The total SGRQ score and the score for each domain range from 0 to 100, with higher scores indicating worse HRQoL.
  Change from baseline defined as: post baseline - baseline value. Mixed model analysis with fixed effects of visit, GAPBSL stage, FVCBSL (cut off <70%), DLCOBSL (cut off <40%), number of comorbidities and baseline score by visit interaction.
Time Frame: At baseline and at 3 months.
Population: Treated Set (TS): all patients who were enrolled in the trial and have received at least once nintedanib during the trial. Any analysis on primary, secondary and safety endpoints was performed in the TS. The number of participants analysed displays the number of participants with available data at the timepoint of interest, at 3 months.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Nintedanib for Patients With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 180
Score on a scale
  total score: number analyzed (Participants) | 160
  total score | 2.08 [-2.15 to 6.31]
  symptoms domain score: number analyzed (Participants) | 160
  symptoms domain score | -2.31 [-5.89 to 1.27]
  activity domain score: number analyzed (Participants) | 160
  activity domain score | 3.37 [-1.15 to 7.89]
  psychosocial impact domain score: number analyzed (Participants) | 160
  psychosocial impact domain score | 2.88 [-2.1 to 7.85]

2. Secondary Outcome: Mean Change From Baseline of Dyspnoea Burden With Modified Medical Research Council Scale (mMRC) Score
Description: The modified Medical Research Council (mMRC) consists of a 5-level rating scale (grades 0-4) based on the patient's perception of dyspnoea (perception of breathlessness) in daily activities, with grade 4 representing the most severe category.
  Change from baseline defined as: post baseline - baseline value. Mixed model analysis with fixed effects of visit, GAPBSL stage, FVCBSL (cut off <70%), DLCOBSL (cut off <40%), number of comorbidities and baseline score by visit interaction.
Time Frame: At baseline and at 3, 6, 9, and 12 months.
Population: Treated Set (TS): all patients who were enrolled in the trial and have received at least once nintedanib during the trial. Any analysis on primary, secondary and safety endpoints was performed in the TS. The number of participants analysed displays the number of participants with available data at the timepoint of interest.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale.
Arm/Group | Nintedanib for Patients With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 180
Score on a scale.
  At 3 months: number analyzed (Participants) | 160
  At 3 months | 0.30 [0.09 to 0.51]
  At 6 months: number analyzed (Participants) | 160
  At 6 months | 0.31 [0.10 to 0.51]
  At 9 months: number analyzed (Participants) | 160
  At 9 months | 0.40 [0.19 to 0.61]
  At 12 months: number analyzed (Participants) | 160
  At 12 months | 0.39 [0.18 to 0.60]

3. Secondary Outcome: Mean Change Form Baseline to the Follow up Period of Cough Burden With Cough-Visual Analogue Scale (Cough-VAS)
Description: Patients were asked at each study visit to rate their perceived intensity of cough due to their IPF on a vertical VAS ranging from 0 to 100, with endpoints labelled as 'no cough' ('100'), 'moderate cough' ('50'), and 'intense cough' ('0').
  Change from baseline defined as: post baseline - baseline value. Mixed model analysis with fixed effects of visit, GAPBSL stage, FVCBSL (cut off <70%), DLCOBSL (cut off <40%), number of comorbidities and baseline score by visit interaction.
Time Frame: At baseline, and at 3, 6, 9, and 12 months.
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale.
Arm/Group | Nintedanib for Patients With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 180
Score on a scale.
  At 3 months: number analyzed (Participants) | 160
  At 3 months | -0.72 [-4.87 to 3.42]
  At 6 months: number analyzed (Participants) | 160
  At 6 months | -3.73 [-7.92 to 0.45]
  At 9 months: number analyzed (Participants) | 160
  At 9 months | -2.13 [-6.36 to 2.09]
  At 12 months: number analyzed (Participants) | 160
  At 12 months | -1.25 [-5.48 to 2.98]

4. Secondary Outcome: Percentage of Adhered Patients to Nintedanib Treatment With Simplified Medication Adherence Questionnaire (SMAQ)
Description: SMAQ consisted of 6 items of which, four were dichotomous (Yes/No), one was Likert-type and one was an open question. A patient was considered as non-adherent, if he/she gave a positive response to any of the qualitative questions, and in terms of quantification, if the patient had lost one of the two daily doses for more than 2 days or had not taken medication for more than four complete days during the past 3 months.
Time Frame: At 3, 6, 9, and 12 months.
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Nintedanib for Patients With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 180
Percentage of participants
  At 3 months: number analyzed (Participants) | 147
  At 3 months | 70.75
  At 6 months: number analyzed (Participants) | 143
  At 6 months | 74.13
  At 9 months: number analyzed (Participants) | 141
  At 9 months | 75.18
  At 12 months: number analyzed (Participants) | 138
  At 12 months | 76.81

5. Secondary Outcome: Mean Change of Anxiety in IPF Patients Treated With Nintedanib From Baseline to Follow up Period Via Generalized Anxiety Disorder Screener (GAD-7) Questionnaire
Description: Generalized Anxiety Disorder Screener (GAD-7) is a 7-item instrument validated for anxiety evaluation that could be used in an outpatient setting. Patients were asked at all study visits to indicate how often they experienced anxiety symptoms over the previous two weeks on a 4-point Likert scale as follows: 0 = 'not at all'; 1 = 'several days'; 2 = 'more than half the days'; and 3 = 'nearly every day'.
  Change from baseline defined as: post baseline - baseline value. Mixed model analysis with fixed effects of visit, GAPBSL stage, FVCBSL (cut off <70%), DLCOBSL (cut off <40%), number of comorbidities and baseline score by visit interaction.
Time Frame: At baseline, and at 3, 6, 9, and 12 months.
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale.
Arm/Group | Nintedanib for Patients With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 180
Score on a scale.
  At 3 months: number analyzed (Participants) | 160
  At 3 months | 0.09 [-1.19 to 1.38]
  At 6 months: number analyzed (Participants) | 160
  At 6 months | 0.48 [-0.81 to 1.77]
  At 9 months: number analyzed (Participants) | 160
  At 9 months | 0.77 [-0.53 to 2.07]
  At 12 months: number analyzed (Participants) | 160
  At 12 months | 0.97 [-0.33 to 2.26]

6. Secondary Outcome: Percentage of Patients That Use Long Term Oxygen Treatment (LTOT)
Description: Percentage of patients that use Long Term Oxygen Treatment (LTOT) is presented.
Time Frame: At baseline, and at 3, 6, 9, and 12 months.
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Nintedanib for Patients With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 180
Percentage of participants
  At baseline | 17.78
  At 3 months: number analyzed (Participants) | 165
  At 3 months | 16.97
  At 6 months: number analyzed (Participants) | 153
  At 6 months | 16.34
  At 9 months: number analyzed (Participants) | 150
  At 9 months | 15.33
  At 12 months: number analyzed (Participants) | 149
  At 12 months | 15.44

7. Primary Outcome: Mean Change From Baseline in Health Related Quality of Life (HRQoL) Using SGRQ Score at 6 Months
Description: as for outcome 1
Time Frame: At baseline and at 6 months.
Population: Treated Set (TS): all patients who were enrolled in the trial and have received at least once nintedanib during the trial. Any analysis on primary, secondary and safety endpoints was performed in the TS. The number of participants analysed displays the number of participants with available data at the timepoint of interest, at 6 months.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Nintedanib for Patients With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 180
Score on a scale
  total score: number analyzed (Participants) | 160
  total score | 3.55 [-0.71 to 7.8]
  symptoms domain score: number analyzed (Participants) | 160
  symptoms domain score | -1.28 [-4.9 to 2.33]
  activity domain score: number analyzed (Participants) | 160
  activity domain score | 4.18 [-0.37 to 8.73]
  psychosocial impact domain score: number analyzed (Participants) | 160
  psychosocial impact domain score | 4.76 [-0.25 to 9.77]

8. Primary Outcome: Mean Change From Baseline in Health Related Quality of Life (HRQoL) Using SGRQ Score at 9 Months
Description: as for outcome 1
Time Frame: At baseline and at 9 months.
Population: Treated Set (TS): all patients who were enrolled in the trial and have received at least once nintedanib during the trial. Any analysis on primary, secondary and safety endpoints was performed in the TS. The number of participants analysed displays the number of participants with available data at the timepoint of interest, at 9 months.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Nintedanib for Patients With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 180
Score on a scale
  total score: number analyzed (Participants) | 160
  total score | 4.64 [0.36 to 8.92]
  symptoms domain score: number analyzed (Participants) | 160
  symptoms domain score | -1.07 [-4.72 to 2.57]
  activity domain score: number analyzed (Participants) | 160
  activity domain score | 5.36 [0.78 to 9.94]
  psychosocial impact domain score: number analyzed (Participants) | 160
  psychosocial impact domain score | 6.09 [1.05 to 11.13]

9. Primary Outcome: Mean Change From Baseline in Health Related Quality of Life (HRQoL) Using SGRQ Score at 12 Months
Description: as for outcome 1
Time Frame: At baseline and at 12 months.
Population: Treated Set (TS): all patients who were enrolled in the trial and have received at least once nintedanib during the trial. Any analysis on primary, secondary and safety endpoints was performed in the TS. The number of participants analysed displays the number of participants with available data at the timepoint of interest, at 12 months.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Nintedanib for Patients With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 180
Score on a scale
  total score: number analyzed (Participants) | 160
  total score | 6.00 [1.72 to 10.28]
  symptoms domain score: number analyzed (Participants) | 160
  symptoms domain score | -1.03 [-4.67 to 2.62]
  activity domain score: number analyzed (Participants) | 160
  activity domain score | 6.19 [1.61 to 10.77]
  psychosocial impact domain score: number analyzed (Participants) | 160
  psychosocial impact domain score | 8.17 [3.13 to 13.22]

ADVERSE EVENTS:
Time Frame: Up to 52 weeks.
Description: Treated Set (TS): all patients who were enrolled in the trial and have received at least once nintedanib during the trial. Any analysis on primary, secondary and safety endpoints was performed in the TS.
Arm/Group | Nintedanib for Patients With Idiopathic Pulmonary Fibrosis
All-Cause Mortality (participants affected / at risk) | 8/180
Serious Adverse Events (participants affected / at risk) | 10/180
Other Adverse Events (participants affected / at risk) | 12/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib for Patients With Idiopathic Pulmonary Fibrosis (N=180)
Cardiac arrest (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
COVID-19 (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ischaemic stroke (Nervous system disorders) | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Disease progression (General disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib for Patients With Idiopathic Pulmonary Fibrosis (N=180)
Diarrhoea (Gastrointestinal disorders) | 12

LIMITATIONS AND CAVEATS:
Study is characterized by inherent limitations attributed to its non-interventional nature. Given that idiopathic pulmonary fibrosis (IPF) diagnosis was done by treating physician, substantial variability in diagnosis may exist. As patient reported outcomes (PROs) were utilized to evaluate, it is important to be aware of potential bias related to such subjective measures. Given the small numbers and heterogeneous population no comparisons / causal associations could be assessed in study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT03710824/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT03710824/SAP_001.pdf